CLINICAL TRIAL: NCT02236793
Title: Phase III, Multicentre, Randomized, Parallel Group, Double Blinded and Control Group Clinical Trial to Assess the Effectiveness of BioChaperone PDGF-BB In the Treatment of Chronic Diabetic Foot Ulcer
Brief Title: A Phase 3 Clinical Trial to Assess the Effectiveness of BioChaperone PDGF-BB In the Treatment of Chronic Diabetic Foot Ulcer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adocia (Industry)
Collaborators: Virchow Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BC1-CT4
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BioChaperone PDGF-BB (Experimental): BioChaperone PDGF-BB administered every other day at the dose of 4µg/cm² for 20 weeks or until wound closure, associated with Standard of Care
  Interventions: Drug: BioChaperone PDGF-BB
- Standard of Care (Placebo Comparator): Normal saline solution applied every other day at the same volume for up to 20 weeks, associated with standard wound care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: BioChaperone PDGF-BB
  Arms: BioChaperone PDGF-BB
Other: Standard of Care
  Arms: Standard of Care

SUMMARY:
The present clinical trial is designed to assess the effectiveness of BioChaperone PDGF-BB applied at 4 µg/cm² every other day for up to 20 weeks and associated to Standard of Care as compared to Standard of Care alone for the treatment of neuropathic and neurovascular diabetic foot ulcers.(In order to ensure the double-blinding of the treatments, a sterile normal saline solution presented in the same multi-dose spray vials than BioChaperone PDGF-BB will be applied on patients of the control group).

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years old or older, with type 1 or 2 diabetes mellitus
* Patient with a single ulcer on the treated feet
* Patient able and willing to provide informed consent
* Patient able and willing to comply with protocol visits and procedure
* Patient willing to use an off-loading method during the whole duration of the study
* Full-thickness plantar, lateral or dorsal ulcer of the extremity (below the malleolus), excluding inter-digits ulcer (web spaces), extending through the epidermis and dermis, but not involving bone, tendons, ligaments or muscles (grade IA as defined by University of Texas Diabetic Wound Classification or Grade 1 according to Wagner classification)
* Chronic ulcer of at least six weeks despite appropriate wound care
* Ulcer area measured with the formula Length x Width x 0.8 following sharp debridement, of 1 to 10 cm², both inclusive
* Well controlled infection or cellulitis (systemic antibiotherapy) before Baseline Visit
* Peripheral neuropathy as assessed by Semmes- Weinstein monofilament test or by the bio esthesimeter (vibration perception threshold).
* Ankle brachial pressure index > 0.60 and <1.3
* Women surgically sterile, post-menopausal, or agree to practice adequate contraception and have a negative pregnancy test at screening. Non-nursing

Exclusion Criteria:

* Inter digit ulcers
* Ulcer of other cause or origin: electrical, chemical or radiation insult, bedsores, vascular ulcer or Charcot deformities ulcers
* Charcot foot.
* Wound originated from amputation bed
* Active ulcer infection assessed by clinical examination and radiography if necessary. Presence of necrosis, purulence or sinus tracts that cannot be removed by debridement and controlled by standard wound care.
* Active osteomyelitis affecting the area of the target ulcer
* Poorly controlled diabetes (uncontrolled glycemia: HbA1c% >= 10%), renal failure (serum creatinine > 3.0 mg/dL), poor nutritional status (albumin < 3.0 g/dL or total protein < 6.5 g/dL)
* Known connective tissue or malignant disease
* Concomitant treatment with corticosteroids, immunosuppressive agents, radiation therapy, or anticancer chemotherapy
* Use of investigational drug/device or growth factor within 30 days
* Topical application of any advance wound care on this wound (antiseptics, antibiotics, debriders, enzyme) within 7 days
* Vascular reconstruction within 8 weeks
* Patients expected to be noncompliant with the protocol (not available for the duration of the trial, treatment or wound care compliance), or felt to be unsuitable by the Investigator for any other reason.
* A history of severe cerebrovascular events

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Incidence of complete wound closure. | 20 weeks

SECONDARY OUTCOMES:
Time to achieve complete wound closure. | 20 weeks
Percentage reduction in total ulcer surface area at each visit. | 20 weeks
Incidence of complete wound healing | 10 weeks
Number of ulcer recurrence observed 12 weeks after wound healing. | 32 weeks
Treatment emergent adverse events. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arun Bal, MD, Principal Investigator — SL Raheja Hospital
Locations (32):
- India (32):
  - Mediciti Hospital, Hyderabad, Andhra Pradesh
  - SL Raheja Hospital, Mumbai, Maharashtra
  - M.V. Hospital for Diabetes (P) Ltd, Chennai, Tamil Nadu
  - Dr V. Seshiah Diabetes Research Institute, Dr Balaji Diabetes Care centre, Chennai, Taminadu
  - B.J. Medical College and Civil Hospital, Ahmedabad
  - Dr Jivraj Mehta Smarak Health Foundation, Ahmedabad
  - Sangini Hospital, Ahmedabad
  - V.S. General Hospital & Sml NHL Municipal Medical College Sheth, Ahmedabad
  - Rajiv Gandhi Centre for Diabetes and Endocrinology, Aligarh
  - Govt Medical College and Hospital, Chandigarh
  - Sri Ramachandra Medial Centre, Chennai
  - The Madras Diabetes Research Foundation, Chennai
  - The Madras Medical Mission, Chennai
  - Gandhi Medical College & Hospital, Hyderabad
  - Nizam's Institute of Medical Sciences, Hyderabad
  - Sumana Hospital, Hyderabad
  - Surakshaka diabetic Centre(P) Ltd, Hyderabad
  - SMS Medical College & Attached Hospital, Jaipur
  - ILS Hospital, Kolkata
  - IPGME & R and SSKM Hospital, Kolkata
  - Nightingale Hospital, Kolkata
  - Rabindranath Tagore International Insitute of cardiac Sciences, Kolkata
  - Fortis Hospital Phase, Mohali
  - Seth G.S. Medical College and K.E.M Hospital, Mumbai
  - Mysore Medical College & Research Institute, Mysore
  - Govt Medical college & Hospital Medical Square, Nagpur
  - Indira Gandhi Govt Medical College and Hospital, Nagpur
  - B.J. Govt. Medical College and Sassoon Hospital, Pune
  - Inamdar Multispeciality Hospital, Pune
  - Poona Hospital & Research Centre, Pune
  - Shree Giriraj Multispeciality Hospital, Rajkot
  - King Georges Hospital, Visakhapatnam